CLINICAL TRIAL: NCT02401165
Title: Quantification of GADD34 Expression in Rheumatoid Arthritis
Brief Title: Quantification of GADD34 Expression in RA
Acronym: GADD34-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012-A01416-37
Record Dates: First submitted 2015-03-24; First posted 2015-03-27 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Rheumatoid Arthritis
Keywords: GADD34; Unfolded Protein Response; Anti-citrullinated protein antibodies
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Hematologic Tests

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- patient (Other): patient
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — blood test

SUMMARY:
GADD34 is an inducible cofactor of protein phosphatase 1, which has an important role in the Unfolded Protein Response (UPR). UPR is a cellular response to ER stress which is implicated in several autoimmune diseases. GADD34 has been shown to be necessary for proinflammatory cytokine production in response to viral infection in murine models. Nevertheless, the role of GADD34 in cytokine production in humans remains to be elucidated. Here, we investigate the interest of GADD34 in rheumatoid arthritis (RA), in which proinflammatory cytokines have an important pathogenic role.

A case-control study on GADD34 gene expression in PBMC of patients (n=75) with RA and age- and sex-matched healthy controls (n=25). GADD34 gene expression levels in PBMC were measured by quantitative PCR.

DETAILED DESCRIPTION:
The endoplasmic reticulum (ER) is the subcellular compartment where transmembrane and secreted proteins are produced. In normal conditions biosynthesis rate, folding and trafficking of the proteins are tightly regulated through an efficient 'quality control' system. The ER responds to the accumulation of misfolded proteins in its lumen through different signaling pathways known as the unfolded protein response (UPR) [1]. Upon activation, the ER transmembrane protein PERK phosphorylates the alpha subunit of the eukaryotic initiation factor eIF2 [2]. Under these conditions, the transcription factor ATF4 directs the expression of genes involved in resistance to oxidative stress, in amino acid metabolism, as well as the expression of GADD34 (Growth arrest and DNA damage-inducible gene 34) [3]. GADD34 is a regulatory subunit of PP1 phosphatase which dephosphorylates eIF2alpha [4], representing a negative feedback loop of UPR, essential for protein synthesis recovery and cell survival [5].

The UPR is more than just an adaptive response to unfolded protein accumulation in the ER, and UPR signaling pathways intersect with immune responses at many levels [6]. In B lymphocytes activation of UPR is part of the normal program of cell differentiation, playing an important role in immunoglobulin synthesis [7]. ER stress has also been implicated in the pathogenesis of many human diseases, including metabolic, neurodegenerative diseases, and cancer [8]. A direct link between UPR and inflammation has been demonstrated for the development of autoimmune diseases such as inflammatory bowel disease [9].

Rheumatoid arthritis is a chronic multifactorial inflammatory disease. Proinflammatory cytokines, such as TNF-alpha and IL-6, secreted by macrophages and monocytes have an important pathogenic role in the phases of inflammation, synovial proliferation and cartilage damage [10]. Rheumatoid factor (RF) has been the most widely used antibody to diagnose RA [11]; anti-citrullinated protein antibodies (ACPA) have also been included in the diagnostic criteria of ACR/EULAR in 2010 [12] and they are highly associated with the development of erosive RA [13].

GADD34 has recently been shown to be necessary for the production of proinflammatory cytokines by dendritic cells and fibroblasts exposed to double-strand RNA in a murine model [14]. In fibroblasts, GADD34 expression is dependent on PKR (Protein Kinase RNA-activated) activation, showing a direct link between pathogen detection and the eIF2alphaP/ATF4 pathway of UPR. The importance of this link for anti-viral immunity has been demonstrated by the mortality of GADD34-deficient neonate mice infected by Chikungunya virus, due to a significant reduction of IFN-beta production [15]. It has been proposed that GADD34 could have a qualitative role on the selection of mRNAs being translated in particular conditions, such as viral infections [16]. These results suggest that GADD34 might be a key molecule of inflammatory processes in human pathologies as well; however, the role of GADD34 in cytokine production in humans remains to be elucidated. The aim of our study was to investigate GADD34 expression in RA patients.

1. Hetz, C., et al., The unfolded protein response: integrating stress signals through the stress sensor IRE1alpha. Physiol Rev. 91 (4): p. 1219-43.
2. Harding, H.P., et al., Perk is essential for translational regulation and cell survival during the unfolded protein response. Mol Cell, 2000. 5 (5): p. 897-904.
3. Harding, H.P., et al., An integrated stress response regulates amino acid metabolism and resistance to oxidative stress. Mol Cell, 2003. 11 (3): p. 619-33.
4. Novoa, I., et al., Feedback inhibition of the unfolded protein response by GADD34-mediated dephosphorylation of eIF2alpha. J Cell Biol, 2001. 153 (5): p. 1011-22.
5. Novoa, I., et al., Stress-induced gene expression requires programmed recovery from translational repression. Embo J, 2003. 22 (5): p. 1180-7.
6. Janssens, S., B. Pulendran, and B.N. Lambrecht, Emerging functions of the unfolded protein response in immunity. Nat Immunol. 15 (10): p. 910-919.
7. Iwakoshi, N.N., et al., Plasma cell differentiation and the unfolded protein response intersect at the transcription factor XBP-1. Nat Immunol, 2003. 4 (4): p. 321-9.
8. Wang, S. and R.J. Kaufman, The impact of the unfolded protein response on human disease. J Cell Biol. 197 (7): p. 857-67.
9. Kaser, A., et al., XBP1 links ER stress to intestinal inflammation and confers genetic risk for human inflammatory bowel disease. Cell, 2008. 134 (5): p. 743-56.
10. McInnes, I.B. and G. Schett, The pathogenesis of rheumatoid arthritis. N Engl J Med. 365 (23): p. 2205-19.
11. Ingegnoli, F., R. Castelli, and R. Gualtierotti, Rheumatoid factors: clinical applications. Dis Markers. 35 (6): p. 727-34.
12. Aletaha, D., et al., 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 62 (9): p. 2569-81.
13. Majka, D.S., et al., Duration of preclinical rheumatoid arthritis-related autoantibody positivity increases in subjects with older age at time of disease diagnosis. Ann Rheum Dis, 2008. 67 (6): p. 801-7.
14. Clavarino, G., et al., Protein phosphatase 1 subunit Ppp1r15a/GADD34 regulates cytokine production in polyinosinic:polycytidylic acid-stimulated dendritic cells. Proc Natl Acad Sci U S A. 109 (8): p. 3006-11.
15. Clavarino, G., et al., Induction of GADD34 is necessary for dsRNA-dependent interferon-beta production and participates in the control of Chikungunya virus infection. PLoS Pathog. 8 (5): p. e1002708.
16. Claudio, N., et al., Mapping the crossroads of immune activation and cellular stress response pathways. Embo J. 32 (9): p. 1214-24.

ELIGIBILITY:
Inclusion Criteria:

* patients with rheumatoid arthritis fulfilling the American College of Rheumatology 1987 revised criteria for the classification of RA
* age between 18 and 75
* patients benefiting of social security
* Informed consent signed by the patients

  3 groups of patients were included: patients with DAS28<2.6 (n=25); patients with DAS28>2.6 and<5.1 (n=25): patients with DAS28>5.1 (n=25).

Exclusion Criteria:

* patients not fulfilling inclusion criteria
* patients who receive treatments for other pathologies
* persons protected by the law L1121-5 to L1121-8 of CSP (for example: pregnant women)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
To determine if GADD34 gene expression level in the PBMC of rheumatoid arthritis patients is increased compared to its expression in the PBMC of healthy controls. | 3 years
  GADD34 gene expression level is quantified in the PBMC by quantitative PCR.

SECONDARY OUTCOMES:
To verify the repeatability and reproducibility of GADD34 gene expression quantification by quantitative PCR. | 3 years
  GADD34 transcrit amplification in a sample from a healthy donor and a sample from a patient was measured 25 times in the same experiment in order to assess repeatability and in triplicate in each qPCR experiment (at least 7) in order to assess reproducibility.
To compare GADD34 gene expression level in the PBMC of 3 groups of patients: patients with DAS28<2.6 (low RA activity), DAS28>2.6 and <5.1 (intermediate RA activity), DAS28>5.1 (high RA activity). | 3 years
  GADD34 gene expression level was quantified in the PBMC of the three groups of patients and compared between the three groups.
GADD34 gene expression in synovial cells. | 3 years
  In patients treated with therapeutical arthrocentesis, to compare GADD34 gene expression level in synovial cells compared with its level in PBMC.
GADD34 and cytokine production. | 3 years
  Quantification of Th1 and Th2 cytokines in RA patients serum by luminex technology.

REFERENCES:
- [Derived] Clavarino G, Adriouach S, Quesada JL, Clay M, Chevreau M, Trocme C, Grange L, Gaudin P, Gatti E, Pierre P, Cesbron JY, Dumestre-Perard C. Unfolded protein response gene GADD34 is overexpressed in rheumatoid arthritis and related to the presence of circulating anti-citrullinated protein antibodies. Autoimmunity. 2016;49(3):172-8. doi: 10.3109/08916934.2016.1138220. Epub 2016 Feb 1. PMID 26829377